CLINICAL TRIAL: NCT02001090
Title: Vascular Function on the First Day After Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: REK nr 2013/1758
Record Dates: First submitted 2013-11-27; First posted 2013-12-04 (Estimated); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Coronary Artery Disease
Keywords: Cardiac Surgical Procedures; Heart-Lung Machine; Coronary Artery Bypass; Brachial Artery; Vasodilation; Regional Blood Flow; Ultrasonography
MeSH Terms: conditions — Coronary Artery Disease; Aneurysm

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CABG patients: Patients undergoing cardiac surgery for coronary artery disease with the use of heart-lung machine in St Olavs Hospital Trondheim University Hospital.

SUMMARY:
This study examines the flow mediated dilation (FMD) of the brachial artery before and after cardiac surgery. FMD is measured with ultrasound technique. Increased flow is achieved trough obstructing blood flow with a cuff around the forearm for five minutes. FMD is measured before surgery and on the first morning after the operation.

ELIGIBILITY:
Inclusion Criteria:

* admitted for coronary artery bypass surgery

Exclusion Criteria:

* Ongoing treatment with nitrates or RAAS inhibiting drugs
* unstable coronary syndrome
* unstable circulation/shock
* renal failure
* hepatic failure
* autoimmune or inflammatory disease
* untreated hypertension.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing coronary artery bypass surgery.
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2014-04-29 (Actual); Study Completion 2014-04-29 (Actual)

PRIMARY OUTCOMES:
flow mediated dilation of the brachial artery | one day
  Transitory change in FMD as a consequence of cardiac surgery with use of extra corporal circulation.

SECONDARY OUTCOMES:
Reactive hyperemia | one day
  Transitory change in reactive hyperemia after five minutes of occlusion of forearm blood flow as a consequence of cardiac surgery with the use of extra corporal circulation.

CONTACTS AND LOCATIONS:
Overall Officials: Idar Kirkeby-Garstad, Md. PhD., Study Director — Department of Cardiothoracic Anesthesiolgy and Intensive Care, St. Olav's Hospital, Trondheim, Norway
Locations (1):
- St. Olavs Hospital, Trondheim, Sør Trøndelag, Norway

REFERENCES:
- [Result] Dedichen HH, Hisdal J, Skogvoll E, Aadahl P, Kirkeby-Garstad I. Reduced reactive hyperemia may explain impaired flow-mediated dilation after on-pump cardiac surgery. Physiol Rep. 2017 May;5(10):e13274. doi: 10.14814/phy2.13274. PMID 28554963